CLINICAL TRIAL: NCT02441166
Title: Evaluation of the Diagnostic Value of Level of Bone Marrow Tryptase in Adult Systemic Mastocytosis
Brief Title: Diagnostic Value of Bone Marrow Tryptase in Systemic Mastocytosis
Acronym: EvaTryMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/14/7387; 2015-A00351-48 (Other: Id-RCB number)
Record Dates: First submitted 2015-05-05; First posted 2015-05-12 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Systemic Mastocytosis
Keywords: Bone marrow tryptase; cutaneous mastocytosis
MeSH Terms: conditions — Mastocytosis, Systemic; Mastocytosis, Cutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mastocytosis diagnosis (Other): For each enrolled subject, 5 mL sample of peripheral blood and 1 mL sample of BM aspirate will be collected the same day to do diagnosis mastocytosis tests (quantification of the kit mutations by qPCR, plasma tryptase level, immunophenotyping of BM mastocytes by flow cytometry, BM tryptase level, degree of dilution of the BM aspirate...) using the WHO criteria as the reference standard.
  Interventions: Procedure: Mastocytosis diagnosis

INTERVENTIONS:
Procedure: Mastocytosis diagnosis — Some samples will be extracted from bone marrow aspirate and peripheral blood on the inclusion day to do diagnosis tests. WHO criteria will be used as the reference standard.

SUMMARY:
The hypothesis of the study is that Bone Marrow Tryptase (MT) level is a diagnostic marker of Systemic Mastocytosis (SM). Determination of the bone marrow tryptase in Bone Marrow Aspirate (BMA) could be a new diagnostic criteria for systemic mastocytosis with sensitivity close to 100% and a low false negative rate. This new test could be useful to improve the ability to diagnose accurately systemic mastocytosis (in particular the indolent forms). Because of its limited invasiveness compared to bone marrow biopsy, it could also be considered as a test performed before bone marrow biopsy. Only patients with high bone marrow tryptase would then undergo bone marrow biopsy.

In the future and if validated by this study, bone marrow tryptase could be a useful marker of mast cell load and help to monitor the efficacy of treatment in systemic mastocytosis.

DETAILED DESCRIPTION:
Mastocytosis are a group of disorders characterized by clonal accumulation of mast cells in various organs. Diagnosis of mastocytosis is challenging and patients remain undiagnosed for years. Using the diagnostic criteria defined by the World Health Organization (WHO) mastocytosis can be divided between Cutaneous Mastocytosis (CM) and Systemic Mastocytosis (SM).

Study suggested that measurement of tryptase in plasma from a Bone Marrow Aspirate (from BMA) could be useful for the diagnosis of SM. Results from a preliminary study at Toulouse University Hospital suggested that a Bone Marrow Tryptase Level (MT) of 50 µg/L or more may be a more sensitive diagnostic criterion (sensitivity of 94.7%) than the histological result of BMB (the major diagnostic criterion for SM with a sensitivity of 68 to 80% in expert centers) for diagnosis of SM in patients with mastocytosis in skin.

Because this preliminary study was done on a limited number of patients and in a single center, the diagnostic value of MT for the diagnosis of SM, has to be confirmed on a larger and more representative population.

In addition, the investigators propose to evaluate:

* The diagnostic accuracy of MT for diagnosis of SM in patients without mastocytosis in skin;
* The diagnostic accuracy of absolute and corrected MT for diagnosis of SM with and without mastocytosis in skin;
* The diagnostic accuracy of MT/ST ratio for diagnosis of SM with and without mastocytosis in skin;
* The diagnostic accuracy of flow cytometry performed on cells collected by BMA and maintained in a preservative solution for diagnosis of SM with and without mastocytosis in skin;
* The diagnostic accuracy of quantification of the fraction of KIT mutation-positive cells in peripheral blood for diagnosis of SM with and without mastocytosis in skin;
* Correlation the results of quantification of the fraction of KIT mutation-positive cells in peripheral blood with results of MT level, results of MT/ST ratio and results of absolute and corrected MT;
* Correlation the results of the CF performed both on the EDTA/TransFix® tubes and on sodium heparin tubes and validate the transport conditions (20-25°C within 24 to 96H) for the CF; these analyzes will be performed on the first 50 samples of BMA.

The samples for these diagnosis tests will be made on the day of inclusion. For each enrolled patient, one 5 mL sample of peripheral blood (EDTA) and 1 mL samples of BM aspirate (0,5 mL in a EDTA/TransFix® tube et 0,5 mL in a sodium heparinate tube) will be collected the same day, and shipped in less than 24 to 96H (+20-25°C) to a central laboratory.

For each patient, genomic DNA from total leucocytes will be purified from the peripheral blood EDTA samples, and used later for the quantification of the kit mutations by real-time qPCR. The plasma tryptase level will be measured from the peripheral blood EDTA sample after an aliquot has been taken for DNA extraction. The bone marrow aspirate sample will be used first for immunophenotyping of BM mastocytes by flow cytometry (FC), and then, after centrifugation, for measurement of BM tryptase level. The degree of dilution of the BM aspirate by peripheral blood will be estimated by comparing the percentage of CD16bright vs. CD16low granulocytes in BM samples, and used to adjust the BM tryptase. Tryptase measurements will be made from EDTA or Na, heparinate plasma, using a standardized fluoro enzyme immunoassay on an automated analyzer. Immunophenotyping of BM mastocytes will be performed on BM aspiration stabilized by TransFix® (a Cellular Antigen Stabilisation Reagent) (and for firsts 50 samples on BM aspiration in Na, heparinate) using a pre-defined mixture of anti-CD45/CD117/CD34/CD2/CD25/CD16 antibodies, coupled to appropriate fluorochromes. Genomic DNA from BM leucocytes will be extracted from 300-500µL of peripheral blood (both anti coagulated with EDTA) using a Promega DNA automated extractor, and subsequently stored at +4°C. Quantitative PCR will be performed using a pre-validated qPCR assay (Life Technologies, Foster City, CA) with a 7900HT Fast Real-Time PCR System (Life Technologies).

The end of study visit is performed the same day that the patient is seen to be made aware of the results of the clinical and laboratory investigations made. This is also the day when the planned medical management of mastocytosis is discussed.

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of systemic mastocytosis, for whom bone marrow sampling (bone marrow biopsy and/or bone marrow aspiration) is carried out as part of normal workup of the disease in the center of reference and centers of competence in mastocytosis.
* Patient whose written informed consent has been obtained.

Exclusion Criteria:

* Patients with a contra-indication to marrow sampling (anticoagulant and/or anti-clotting treatments,
* Thrombocytopenia < 50 000/mm2) for whom it is impossible to formally conclude the final type of mast cell disease: SM, CM, mast cell activation syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2015-10-06 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Bone marrow tryptase level | Day 4 after bone marrow aspiration
  Aliquot of the bone marrow aspirate sample will be used after centrifugation for measurements of bone marrow tryptase level.

SECONDARY OUTCOMES:
The bone marrow tryptase level for differential diagnosis between systemic mastocytosis and cell mast activation syndrome | Day 4 after bone marrow aspiration
  Aliquot of the bone marrow aspirate sample will be used after centrifugation for measurements of bone marrow tryptase level.
The bone marrow tryptase/serum tryptase ratio for diagnosis of systemic mastocytosis with and without mastocytosis in skin | Day 4 after bone marrow aspiration
The absolute and corrected bone marrow tryptase level for diagnosis of systemic mastocytosis with and without mastocytosis in skin | Day 4 after bone marrow aspiration
  The degree of dilution of the bonne marrow aspirate by peripheral blood will be estimated by comparing the percentage of CD16bright vs CD16low granulocytes in bone marrow samples and used to adjust the bone marrow tryptase.
Flow cytometry performed on cells collected by bone marrow aspirate and maintained in a preservative solution (TransFix®) to detect mast cells expressing CD25 and/or CD2 for diagnosis of systemic mastocytosis with and without mastocytosis in skin | Day 4 after bone marrow aspiration
  Immunophenotyping of bone marrow mastocytes will be performed on bone marrow aspiration stabilized by Transfix using a pre-defined mixture of anti-CD45/CD117/CD34/CD2/CD25/CD16 antibodies.
Quantification of KIT mutations-positive cells fraction in peripheral blood for systemic mastocytosis diagnosis,correlation with results of medullar tryptase level, medullar/systemic tryptase ratio and absolute and corrected medullar tryptase level | Day 4 after bone marrow aspiration
  Genomic DNA from total leucocytes will be purified from the peripheral blood samples and used for the quantification of the kit mutation by qPCR

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Livideanu, MD, Principal Investigator — University Hospital, Toulouse
Locations (8):
- France (7):
  - CHU Bordeaux Hôpital Haut-Lévêque, service de dermatologie, Bordeaux
  - CHU de Caen, service d'hématologie, Caen
  - CHU Dupuytren service d'hématologie, Limoges
  - CHU Lyon Sud, service de médecine interne, Lyon
  - Hôpital Necker, service d'hématologie, Paris
  - Hôpital Pité Salpétrière, Paris
  - CHU Toulouse, Hôpital Larrey, service de dermatologie, Toulouse
- CHU Fort de France, service de dermatologie, Fort-de-France, Martinique

REFERENCES:
- [Background] Valent P, Horny HP, Escribano L, Longley BJ, Li CY, Schwartz LB, Marone G, Nunez R, Akin C, Sotlar K, Sperr WR, Wolff K, Brunning RD, Parwaresch RM, Austen KF, Lennert K, Metcalfe DD, Vardiman JW, Bennett JM. Diagnostic criteria and classification of mastocytosis: a consensus proposal. Leuk Res. 2001 Jul;25(7):603-25. doi: 10.1016/s0145-2126(01)00038-8. PMID 11377686
- [Background] Valent P, Akin C, Escribano L, Fodinger M, Hartmann K, Brockow K, Castells M, Sperr WR, Kluin-Nelemans HC, Hamdy NA, Lortholary O, Robyn J, van Doormaal J, Sotlar K, Hauswirth AW, Arock M, Hermine O, Hellmann A, Triggiani M, Niedoszytko M, Schwartz LB, Orfao A, Horny HP, Metcalfe DD. Standards and standardization in mastocytosis: consensus statements on diagnostics, treatment recommendations and response criteria. Eur J Clin Invest. 2007 Jun;37(6):435-53. doi: 10.1111/j.1365-2362.2007.01807.x. PMID 17537151
- [Background] Akin C, Valent P, Metcalfe DD. Mast cell activation syndrome: Proposed diagnostic criteria. J Allergy Clin Immunol. 2010 Dec;126(6):1099-104.e4. doi: 10.1016/j.jaci.2010.08.035. Epub 2010 Oct 28. PMID 21035176
- [Background] Alvarez-Twose I, Gonzalez de Olano D, Sanchez-Munoz L, Matito A, Esteban-Lopez MI, Vega A, Mateo MB, Alonso Diaz de Durana MD, de la Hoz B, Del Pozo Gil MD, Caballero T, Rosado A, Sanchez Matas I, Teodosio C, Jara-Acevedo M, Mollejo M, Garcia-Montero A, Orfao A, Escribano L. Clinical, biological, and molecular characteristics of clonal mast cell disorders presenting with systemic mast cell activation symptoms. J Allergy Clin Immunol. 2010 Jun;125(6):1269-1278.e2. doi: 10.1016/j.jaci.2010.02.019. PMID 20434205
- [Background] Barete S, Assous N, de Gennes C, Grandpeix C, Feger F, Palmerini F, Dubreuil P, Arock M, Roux C, Launay JM, Fraitag S, Canioni D, Billemont B, Suarez F, Lanternier F, Lortholary O, Hermine O, Frances C. Systemic mastocytosis and bone involvement in a cohort of 75 patients. Ann Rheum Dis. 2010 Oct;69(10):1838-41. doi: 10.1136/ard.2009.124511. Epub 2010 Jun 22. PMID 20570833
- [Background] Paul C, Sans B, Suarez F, Casassus P, Barete S, Lanternier F, Grandpeix-Guyodo C, Dubreuil P, Palmerini F, Mansfield CD, Gineste P, Moussy A, Hermine O, Lortholary O. Masitinib for the treatment of systemic and cutaneous mastocytosis with handicap: a phase 2a study. Am J Hematol. 2010 Dec;85(12):921-5. doi: 10.1002/ajh.21894. PMID 21108325